CLINICAL TRIAL: NCT00847964
Title: SYM-08-001: A Pilot Study to Evaluate the Safety and Feasibility of Algisyl-LVR™ as a Method of Left Ventricular Restoration in Patients With Dilated Cardiomyopathy Undergoing Open-heart Surgery
Brief Title: Safety and Feasibility of Algisyl-LVR™ as a Method of Left Ventricular Restoration in Patients With DCM Undergoing Open-heart Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LoneStar Heart, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYM-08-001
Record Dates: First submitted 2009-02-17; First posted 2009-02-19 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2012-11

CONDITIONS: Dilated Cardiomyopathy
Keywords: Heart Failure
MeSH Terms: conditions — Cardiomyopathy, Dilated; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Algisyl-LVR implants (Experimental): Algisyl-LVR implants to the left ventricular wall
  Interventions: Device: Algisyl-LVR

INTERVENTIONS:
Device: Algisyl-LVR — method of left ventricular restoration in patients with dilated cardiomyopathy

SUMMARY:
This is a pilot study to evaluate the feasibility and safety of the Algisyl-LVR™ device. The purpose of this study is to investigate Algisyl-LVR™ employed as a method of left ventricular restoration in patients with dilated cardiomyopathy who are scheduled to undergo routine open heart surgery. Algisyl-LVR™ will be injected into the myocardium under direct visualization during the surgical procedure. This clinical evaluation is intended to provide the initial evidence of the safety and feasibility of the device as well as the procedure used to deploy the device. The results of the initial trial will also help to establish the utility of various assessments in evaluating and following the effects of the device.

DETAILED DESCRIPTION:
Heart Failure (HF) is a progressive condition that has diverse etiologies with only 50 percent of patients presenting at diagnosis with a defined reason for developing the disease. However, estimates are that over half of all patients presenting with HF have coronary artery disease (CAD) as the primary etiology. The most common etiologies among HF patients without CAD have been reported to be systemic hypertension and valvular disease. Irrespective of the etiology, the majority of patients with HF have symptoms due to an impairment of left ventricular (LV) myocardial function. HF is a progressive condition that results from myocardial damage. This damage can be caused by predisposing conditions or an acute event that leads to cardiac remodeling. The principal manifestation of such progression and cardiac remodeling is a change in the geometry and structure of the left ventricle (LV), such that the chamber dilates and/or hypertrophies and becomes more spherical. The cardiac remodeling is maladaptive and its progression leads to worsening of the clinical symptoms of HF, characterized by limited exercise tolerance and edema. Despite optimal medical management, HF is progressive in nature and patients have a mortality rate of over 50 percent in 5 years.

Structural heart abnormalities are known to play a central role in HF, and clinical evidence supports a strong causal relationship between cardiac chamber dilation and heart failure. Because dilation, and not contractile dysfunction, appears to be responsible for the severity of the disease, the mitigation or prevention of the deleterious dilation process appears to be an important therapeutic target for HF patients. Hence, a therapy that specifically targets progressive LV dilatation and remodeling by reshaping and reducing the LV chamber size may offer an important new alternative in the treatment of HF.

Algisyl-LVR™ is a single use, multiple component device under development for the indication to prevent or reverse the progression of heart failure (HF) by providing implanted space-occupying material in the myocardium to affect LV shape and prevent or reverse LV enlargement. The intended clinical benefits of Algisyl-LVR™ are to improve the failing heart's structure and function with an associated improvement in the patient's clinical status and quality of life. Data from this current study will be used to evaluate the initial feasibility of this novel therapeutic device.

The objective of this pilot study is to evaluate the feasibility and safety of the Algisyl-LVR™ device. No formal hypothesis testing will be performed. Descriptive statistics will be used to summarize operator (surgeon) experience and patient outcomes. The results of the study will be used to assess the design of the device and feasibility of the procedures to use the device. The study will also guide the design and sample size of future studies.

This study will be conducted at a several centers in Europe. The surgeon's experience with the use of the device will be collected and evaluated. Measures of safety and tolerability of Algisyl-LVR™ will be evaluated through analysis of adverse experiences, clinical laboratory tests, electrocardiograms, physical examinations, echocardiographic measures and magnetic resonance imaging (MRI). Measurements at specified time intervals will be compared to baseline values obtained prior to treatment.

Patients will be evaluated prior to the procedure, during the immediate post operative period, and then, return to the clinic at 8 days, 3 months, 6 months, 12 months, 18 months and 24 months after the procedure for follow-up evaluations.

ELIGIBILITY:
Inclusion Criteria

1. The patients must be able and willing to give written informed consent.
2. The patients will be adult (age ≥ 18 years and </= 75 years) males or females who are scheduled to undergo open-chest coronary artery bypass grafting surgery and/or valve repair/replacement.
3. The patients must be on stable, evidence-based therapy for heart failure.
4. The patients will have an ejection fraction equal to or less than 40% and a left ventricular end diastolic dimension indexed to body surface area (LVEDDi) of 30 to 40mm/m2 (LVEDD/BSA).
5. Patients must have symptomatic heart failure with a New York Heart Association (NYHA) class of III or IV
6. If female, the patients must be (a) post-menopausal, (b) surgically sterile, or (c) using adequate birth control and have a negative serum pregnancy test within 7 days prior to administration of study device.

Exclusion Criteria:

1. Emergent open heart surgery or cardiogenic shock.
2. Right-sided heart failure.
3. Patients scheduled to undergo pulmonic or tricuspid valve replacements.
4. Patients who have undergone a previous mid-sternotomy or thoracotomy surgical procedure
5. Patients presenting with a restrictive cardiomyopathy such as due to amyloidosis, sarcoidosis, or hemochromatosis.
6. Patient with a history of constrictive pericarditis.
7. Patients with a Q wave myocardial infarction (MI) within the last 30 days.
8. Patients with a recent history of stroke (within 60 days prior to the surgical procedure)
9. A left ventricular (LV) wall thickness of the LV free-wall, at the mid-ventricular level, of less than 6 mm.
10. Patients with a serum creatinine > 2.0 mg/dL..
11. Clinically significant liver enzyme abnormalities, i.e., AST or ALT more than two times the upper limit of normal and/or bilirubin more than 50% above the upper limit of normal.
12. The patients will not be receiving concurrently an investigational Product in another clinical trial or have received an investigational Product in another clinical trial in the 30 days prior to enrollment.
13. A life expectancy of less than 1 year or any other condition that, in the opinion of the clinical investigator, might compromise any aspect of the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-02; Primary Completion 2011-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Freedom from serious adverse events | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Matschke, MD, Principal Investigator — Heart Center Dresden University Hospital
Locations (3):
- Germany (2):
  - Deutsche Herzzentrum München, München, Bavaria
  - Heart Center of the Technical University of Dresden, Dresden
- John Paul II Hospital, Krakow, Poland